CLINICAL TRIAL: NCT05969132
Title: Fully Digital Guided Gingivectomy in Management of Gummy Smile: Evaluation of Accuracy and Patient Satisfaction
Brief Title: Digital Versus Conventional Guided Gingivectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eslam Hashim, Master Student, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RecIM122209
Record Dates: First submitted 2023-07-22; First posted 2023-08-01 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Altered Passive Eruption of Teeth
Keywords: gummy smile; excessive gingival display; Altered Passive Eruption; gingivectomy; fully digital guided

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The current investigation will be a single-blinded clinical trial. Blinding included the assessor, and the statistician. Its impossible for the operator who performed the surgical procedure to be blinded as the interventions will be completely different and the patient also.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital workflow-based Protocol (Experimental): Fully digital guided gingivectomy procedure
  Interventions: Procedure: Fully digital guided gingivectomy procedure
- Mock-up workflow-based Protocol (Active Comparator): Convectional guided gingivectomy procedure
  Interventions: Procedure: Convectional guided gingivectomy procedure

INTERVENTIONS:
Procedure: Fully digital guided gingivectomy procedure — 1. Full history with clinical and radiographic examination (CBCT) to aid in patient's selection.
  2. Supra- and sub-gingival debridement.
  3. Oral hygiene instructions (OHI)
  4. Presurgical intraoral scanning using an intraoral scanner (IOS)
  5. Fabrication of the Gingivectomy guide:
     * Convert (DICOM) file to STL file then merged to STL file corresponding oral soft tissues 3D data obtained by IOS using software of surgical planning.
     * Digital waxing up with new desired positions of gingival margins and zenith points performed.
     * Designing Gingivectomy guide then exported to a 3D printer and mill a transparent resin gingivectomy guide.
  6. Surgical Procedure: anesthetized the patient using local anesthesia, Surgical incision using 15c blade following CEJ anatomy will be made at each tooth using the Gingivectomy guide as reference to new gingival level and being careful to preserve the gingival papillae without involving the palatal surfaces.
  7. Postoperative care
  Arms: Digital workflow-based Protocol
Procedure: Convectional guided gingivectomy procedure — 1. Full history with clinical and radiographic examination (CBCT) to aid in patient's selection.
  2. Supra- and sub-gingival debridement with OHI
  3. Gingivectomy guide fabrication:
     * Impressions and casts obtained.
     * Waxing-up included new positions of gingival margins and zenith points.
     * Silicone index with condensation silicone impression materials made with pressure on the cast to reproduce the details of the wax, then filled after setting with resin material and placed in the patient's mouth.
     * Resin mock-up trimmed with blade to define the correct new gingival level.
     * After the patient accept the mock-up design will used as Gingivectomy guide.
  4. Surgical Procedure: anesthetized the patient using local anesthesia, Surgical incision using 15c blade following CEJ anatomy will be made at each tooth using the Gingivectomy guide as reference to new gingival level and being careful to preserve the gingival papillae without involving the palatal surfaces.
  5. Postoperative care
  Arms: Mock-up workflow-based Protocol

SUMMARY:
The goal of this randomized controlled clinical study is to compare Fully digital to conventional guided Gingivectomy procedure in management of excessive gingival display caused by altered passive eruption type 1A.

The main question it aims to answer is:

Does the fully digital guided gingivectomy approach able to introduce a more precise, accuracy and reliability technique with more patient satisfaction compared to the conventional guided method?

DETAILED DESCRIPTION:
Nowadays, the concept of smile and dental esthetics is no longer limited to the teeth. The essentials of a smile involve the relationship between the three primary components: the teeth, lip framework, and the gingival scaffold.

The term "pink aesthetics" refers to the aesthetics of gingival tissues, which play a significant influence in smile aesthetics.

Excessive gingival display while smiling, also usually known as a "gummy smile," is a common esthetic concern among dental patients and, being largely viewed as unesthetic, leads many patients to seek some form of treatment to address the issue.

Gummy smile (Excessive gingival display) is recognized by the American Academy of Periodontology (AAP) as a deformity and mucogingival condition that affects the area around the teeth.

This condition could be caused by many etiological factors: short lip, hypermobile/hyperactive lip, short clinical crowns, dentoalveolar extrusion, altered passive eruption (APE), gingival hyperplasia, and vertical maxillary excess.

Altered passive eruption defined as "the gingival margin in the adult is located incisal to the cervical convexity of the crown and removed from the cementoenamel junction of the tooth".

Altered passive eruption classified into two main classes according to the relationship of the gingiva to the anatomic crown and furthermore subdivided those classes according to the position of the osseous crest. The two types are subdivided into four categories: 1A, 1B and 2A, 2B.

The diagnosis of APE is made on a collective clinical and radiographic examination, it begins with analyzing the repose during a natural smile followed by analyzing the gingival display, the alveolar crest level, as well as the lip line of the patient.

Determination can be made whether a gingivectomy alone will suffice or a gingival flap will be needed with or without ostectomy will depend of the diagnosis of APE and classification of each case.

The selection of one technique over another depends on several patient related factors such as esthetics, clinical crown to root ratio, root proximity, root morphology, furcation location, individual tooth position, collective tooth position and ability to restore the teeth.

The gingivectomy approach alone is used when 3 mm gingival tissue or greater exists from bone to gingival crest, and an adequate attached gingiva will remain after surgery (APE type IA).

A diagnostic wax-up then an intraoral fabricated mock-up representing the desired outcome can assist in the selection of proper planning of the need for periodontal surgical approach.

Diagnostic mock-up fabricated using a temporary bis-acrylic resin with a putty guide directly from the wax-up can be used to provide the patient and clinician with an evaluation of the future outcome and can be used as a surgical guide for gingivectomy procedures.

The major limitations with conventional guided gingivectomy procedure would be the time consumed during making and modifying conventional wax-ups as well as the unpredictable estimate of where the gingival margin should be.

Utilization of digital workflows allowed the enhancement of communication and might improve the predictability of contemporary gingivectomy approach.

The introduction of computer-aided design and computer-aided manufacturing (CAD-CAM) techniques has helped surgeons perform more precise and predictable surgery and contributed to improved esthetics.

By combining the use of Digital Smile Design and CAD/CAM technology with (3D) printing, a surgical guide for Gingivectomy procedure could be produced.

The aim of the present study will be to evaluate accuracy and reliability of digital guided method of gingivectomy procedure using CAD CAM technology versus conventional method using resin Mock-up as gingivectomy surgical guide.

Research Question "Does the fully digital guided gingivectomy approach able to introduce a more precise, accuracy and reliability technique with more patient satisfaction compared to the conventional guided method?"

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of Excessive gingival display (3mm or more gingival display at full smiling)
* Patients classified as Altered Passive Eruption Type 1A

Exclusion Criteria:

* Patients need restorative or orthodontic correction.
* Pregnant and lactating females.
* Heavy smoker ≥ 10 cigarettes/day.
* Poor oral hygiene.
* Patients with systemic diseases which could influence the outcome of the therapy e.g.

(Diabetic patients).

* Heavy smoker ≥ 10 cigarettes/day.
* Vulnerable groups of patients e.g. (prisoners, handicapped patients and decisionally impaired individuals)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy of both guides | Immediately postsurgical, 4 weeks and 2 months after surgery
  Intraoral digital scanning for obtaining gingival contour will be made immediately postsurgical, 4 weeks and 2 months after surgery and exported in STL files format.
  Diagnostic waxing-up on poured cast (for group 2) will be digitalized with a model scanner and exported in STL file format.
  Accuracy will be evaluated by:
  * Superimposing postoperative intraoral digital scanning STL files with virtually designed diagnostic waxing STL file (for group 1) and obtain matching differences in height of gingival margin in relation to Muco-gingival junction.
  * Superimposing postoperative intraoral digital scanning STL files with digitized waxing-up STL file (for group 2) and obtain matching differences in height of gingival margin in relation to Muco-gingival junction.

SECONDARY OUTCOMES:
Patient Satisfaction | 2 months
  A 5-item custom made questionnaire will give to the patients to be answered for assessing their satisfaction with the whole procedure and the results of the procedure performed.
  1. Post-operative pain (POP): It will be evaluated indirectly based on the mean consumption (in mg) of analgesics (ibuprofen)* after the surgical procedures (Wessel and Tatakis, 2008).
  2. Post-operative results
  3. Post-operative swelling: It will be reported by the patients through the first week (7 days) postsurgically based on the Verbal Rating Scale (VRS) values (absent, slight, moderate and severe) (García et al., 2008).
  4. Surgery time
  5. Procedure as a whole

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E. Amr, Ass. Prof., Study Director — Faculty of dentistry Ain Shams University
Locations (1):
- Faculty of Fentistry Ain Shams university, Cairo, Egypt

REFERENCES:
- [Background] Ahmed WM, Hans A, Verhaeghe TV, Nguyen C. Managing Excessive Gingival Display Using a Digital Workflow. J Prosthodont. 2020 Jun;29(5):443-447. doi: 10.1111/jopr.13181. Epub 2020 May 6. PMID 32321195
- [Background] Arias DM, Trushkowsky RD, Brea LM, David SB. Treatment of the Patient with Gummy Smile in Conjunction with Digital Smile Approach. Dent Clin North Am. 2015 Jul;59(3):703-16. doi: 10.1016/j.cden.2015.03.007. PMID 26140976
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Bensimon GC. Surgical crown-lengthening procedure to enhance esthetics. Int J Periodontics Restorative Dent. 1999 Aug;19(4):332-41. PMID 10709500
- [Background] Coslet JG, Vanarsdall R, Weisgold A. Diagnosis and classification of delayed passive eruption of the dentogingival junction in the adult. Alpha Omegan. 1977 Dec;70(3):24-8. No abstract available. PMID 276255
- [Background] Davarpanah M, Jansen CE, Vidjak FM, Etienne D, Kebir M, Martinez H. Restorative and periodontal considerations of short clinical crowns. Int J Periodontics Restorative Dent. 1998 Oct;18(5):424-33. PMID 10093519
- [Background] De Rouck T, Eghbali R, Collys K, De Bruyn H, Cosyn J. The gingival biotype revisited: transparency of the periodontal probe through the gingival margin as a method to discriminate thin from thick gingiva. J Clin Periodontol. 2009 May;36(5):428-33. doi: 10.1111/j.1600-051X.2009.01398.x. PMID 19419444
- [Background] Dolt AH 3rd, Robbins JW. Altered passive eruption: an etiology of short clinical crowns. Quintessence Int. 1997 Jun;28(6):363-72. PMID 9477899
- [Background] Dym H, Pierre R 2nd. Diagnosis and Treatment Approaches to a "Gummy Smile". Dent Clin North Am. 2020 Apr;64(2):341-349. doi: 10.1016/j.cden.2019.12.003. Epub 2020 Jan 24. PMID 32111273
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Garber DA, Salama MA. The aesthetic smile: diagnosis and treatment. Periodontol 2000. 1996 Jun;11:18-28. doi: 10.1111/j.1600-0757.1996.tb00179.x. No abstract available. PMID 9567953
- [Background] Garcia B, Larrazabal C, Penarrocha M, Penarrocha M. Pain and swelling in periapical surgery. A literature update. Med Oral Patol Oral Cir Bucal. 2008 Nov 1;13(11):E726-9. PMID 18978715
- [Background] Geevarghese A, Baskaradoss JK, Alsalem M, Aldahash A, Alfayez W, Alduhaimi T, Alehaideb A, Alsammahi O. Perception of general dentists and laypersons towards altered smile aesthetics. J Orthod Sci. 2019 Aug 8;8:14. doi: 10.4103/jos.JOS_103_18. eCollection 2019. PMID 31497573
- [Background] Goldman, H.M. & Cohen, D.W. (1968). Periodontal Therapy. 4ed. St. Louis: C.V. Mosby Company.
- [Background] Gurrea J, Bruguera A. Wax-up and mock-up. A guide for anterior periodontal and restorative treatments. Int J Esthet Dent. 2014 Summer;9(2):146-62. PMID 24765624
- [Background] Herrero F, Scott JB, Maropis PS, Yukna RA. Clinical comparison of desired versus actual amount of surgical crown lengthening. J Periodontol. 1995 Jul;66(7):568-71. doi: 10.1902/jop.1995.66.7.568. PMID 7562348
- [Background] Hejazin, N., Wehbe, C., Wierup, M., Montilla, D.E. & Al-Mashni, L. (2020). Diagnosis and treatment modalities of altered passive eruption: Review and a case report of gummy smile. J Case Rep Images Dent, 6:100034Z07NH2020.
- [Background] Landry, R.G., Turnbull, R.S., & Howley, T. (1988). Effectiveness of benzydamine HCl in the treatment of periodontal post-surgical patients. Res Clin Forum. 10. 105-118.
- [Background] Levine RA. Forced eruption in the esthetic zone. Compend Contin Educ Dent. 1997 Aug;18(8):795-803; quiz 804. PMID 9533338
- [Background] Liu X, Yu J, Zhou J, Tan J. A digitally guided dual technique for both gingival and bone resection during crown lengthening surgery. J Prosthet Dent. 2018 Mar;119(3):345-349. doi: 10.1016/j.prosdent.2017.04.018. Epub 2017 Jul 8. PMID 28689907
- [Background] Patil AS, Ranganath V, Yerawadekar SA, Kumar CN, Sarode GS. Pink Esthetics: A Study on Significant Gingival Parameters. J Contemp Dent Pract. 2020 Feb 1;21(2):207-210. PMID 32381829
- [Background] Pavone AF, Ghassemian M, Verardi S. Gummy Smile and Short Tooth Syndrome--Part 1: Etiopathogenesis, Classification, and Diagnostic Guidelines. Compend Contin Educ Dent. 2016 Feb;37(2):102-7; quiz 108-10. PMID 26905089
- [Background] Perakis N, Cocconi R. The decision-making process in interdisciplinary treatment: digital versus conventional approach. A case presentation. Int J Esthet Dent. 2019;14(2):212-224. PMID 31062001
- [Background] Ruhmann, N.L., Borrasca, C., Araújo, C, A., & Pfau, E.A. (2014). Aesthetic rehabilitation of the "gummy smile" associated to virtual planning with "digital smile design"-DSD. J Surg Clin Dent, 1(1):5-9
- [Background] Simon H, Magne P. Clinically based diagnostic wax-up for optimal esthetics: the diagnostic mock-up. J Calif Dent Assoc. 2008 May;36(5):355-62. PMID 18557126
- [Background] Trushkowsky R, Arias DM, David S. Digital Smile Design concept delineates the final potential result of crown lengthening and porcelain veneers to correct a gummy smile. Int J Esthet Dent. 2016 Autumn;11(3):338-54. PMID 27433549
- [Background] Vercruyssen M, Cox C, Coucke W, Naert I, Jacobs R, Quirynen M. A randomized clinical trial comparing guided implant surgery (bone- or mucosa-supported) with mental navigation or the use of a pilot-drill template. J Clin Periodontol. 2014 Jul;41(7):717-23. doi: 10.1111/jcpe.12231. Epub 2014 Apr 10. PMID 24460748
- [Background] Wessel JR, Tatakis DN. Patient outcomes following subepithelial connective tissue graft and free gingival graft procedures. J Periodontol. 2008 Mar;79(3):425-30. doi: 10.1902/jop.2008.070325. PMID 18315424